CLINICAL TRIAL: NCT01252498
Title: A Pilot Study to Evaluate the Role of Cyclooxygenase Pathway in Radiation Therapy and Chemoradiation Therapy Induced Mucositis in Head and Neck Cancer Patients
Brief Title: Evaluation of the Role of Prostaglandins in Radiation-induced Mucositis
Status: Completed | Type: Observational
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Claire Verschraegen, Professor of Medicine, University of Vermont
Other Study IDs: VCC1005
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Cancer of the Head and Neck; Radiotherapy
Keywords: Cancer of the head and neck; Radiotherapy; Prostaglandins
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Saliva will be collected at 4 time points before, during, immediately after, and several weeks after radiotherapy for head and neck cancer.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Radiotherapy: Patients receiving radiotherapy or chemoradiotherapy for head and neck cancer

SUMMARY:
This study will evaluate the role of cyclooxygenase pathways in radiation-induced and chemoradiation-induced mucositis.

DETAILED DESCRIPTION:
Oral mucositis is a significant toxicity of radiation therapy and chemoradiation therapy in head and neck cancer patients. However the mechanisms that induce such mucositis are not completely understood. Previous work evaluating mucositis in bone marrow transplant patients has suggested that prostaglandin levels may be associated with the appearance of mucositis.

The present study will measure the levels in saliva of the prostaglandins PGE2 and PGI2 before, during, immediately after, and several weeks after radiotherapy for head and neck cancer. These salivary levels will be correlated with clinical observation of mucositis and patient reporting of pain levels.

Improved understanding of the mechanism of mucositis may lead to the development of more effective targeted agents to prevent this problem.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven locoregional Stage 4 squamous cell carcinoma of the oral cavity, larynx, oropharynx or hypopharynx
* Receiving radiation therapy or chemoradiation therapy to the oropharynx
* Older than 18 years old
* ECOG performance status of 0-2
* Life expectancy greater than 2 months
* Signed informed consent

Exclusion Criteria:

* Previous chemotherapy for this malignancy
* Previous radiotherapy to the head and neck
* Other cancer diagnosis within the last 5 years except for non-melanoma skin cancer or non-metastatic prostate cancer
* Patient taking NSAIDs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving radiotherapy or chemoradiotherapy for oral cancers. Consecutive patients will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2010-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Salivary levels of PGE2 and PGI2 during and after radiotherapy | 10 weeks after initiation of therapy

SECONDARY OUTCOMES:
Observed mucositis during and after radiotherapy | 10 weeks after initiation of radiotherapy
Patient reports of oral pain during and after radiation therapy | 10 weeks after initiation of radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Claire Verschraegen, MD, Principal Investigator — University of Vermont/Fletcher Allen Health Care
Locations (1):
- Fletcher Allen Health Care, Burlington, Vermont, United States